CLINICAL TRIAL: NCT04683263
Title: Immediate and Mid-term Effect of a Natural Topical Product in Patients With Musculoskeletal Pain: a Randomized, Double-blinded, and Placebo-controlled Clinical Trial.
Brief Title: Immediate and Mid-term Effect of a Natural Topical Product in Patients With Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uriach Consumer Healthcare (Industry)
Collaborators: Quironsalud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07CRT_VV_323_18-003
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Musculoskeletal Pain; Chronic Pain; Joint Pain; Stiffness of Unspecified Joint, Not Elsewhere Classified
Keywords: Musculoskeletal pain; Chronic pain; Joint mobility; Massage; Rehabilitation
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Arthralgia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blinded and placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients were randomly assigned, using the Excel (Microsoft) RAND function, into 2 groups: treatment group and placebo group, a topical cream with similar characteristics and aspect, without active ingredients. Allocation was concealed from the recruiter and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Fisiocrem®, a topical cream composed of the natural ingredients Arnica montana, Hypericum perforatum, Calendula officinalis, Melaleuca sp. and menthol
  Interventions: Other: Fisiocrem
- Placebo (Placebo Comparator): topical cream with similar characteristics and aspect, without active ingredients.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — topical cream with same composition as Intervention but without active ingredients
  Arms: Placebo
Other: Fisiocrem — a natural topical composition containing Arnica montana, Hypericum perforatum, Calendula officinalis, Melaleuca sp. and menthol
  Arms: Intervention

SUMMARY:
Musculoskeletal pain is a common affection due to ageing, sedentarism and intense exercise practice causing acute and chronic injuries.

The main objective of this trial is to prove efficacy of a natural topical composition containing Arnica montana, Hypericum perforatum, Calendula officinalis, Melaleuca sp. and menthol in pain management in adults with acute or chronic pain.

This randomized, double-blinded and placebo-controlled trial will include 200 patients with musculoskeletal pain, 100 in the intervention group receiving the topical formula and 100 in the placebo group, who will receive a similar formula without active ingredients.

The products will be applied topically twice daily for 14 days in areas with moderate or severe pain.

The study objectives are immediate and long-term pain alleviation, stiffness perception joint mobility, and general recovery perception.

DETAILED DESCRIPTION:
Well-being is understood as the absence of limitations or debilitating conditions that make impossible to enjoy a full and satisfactory life. Among these limitations, a reduced or impaired motility because of painful and inflammatory processes (acute and chronic), can greatly disturb a vital and optimistic attitude.

Chronic pain affects between one-third and one-half of the population only in the UK, and around 20.4% in the US. It is likely to increase with population ageing and tends to be more common in women. Ageing is translated in an increase in the incidence and span of chronic illnesses, including osteoarthritis, fibromyalgia, lower back pain, non-arthritis joint pain or carpal tunnel syndrome, among others. In addition, muscular and joints pain unrelated to any specific disease also tends to appear with age. Beyond that, current lifestyle frequently involves stressful jobs, eventful agendas and non-stop activity either in professional or leisure time. These facts extend the prevalence of chronic pain to younger segments of the population and to people not affected by previous disease.

Sedentary lifestyle and computer-based jobs represent a common cause of muscular contractures and pain, especially in the back and neck areas. Another important contributor to chronic pain is perceived stress and anxiety response systems. As an emergent antagonist phenomenon, increasing awareness of a healthy lifestyle has entailed a rise in the popularity of physical exercise in the last decades. As an example, the number of running events finishers in the U.S. stabilized in 2014 at almost 20 million people, with figures having been on the rise for the previous 25 years. The popularization of exercise programs such as CrossFit illustrate that the trend is directed not only towards a rise in practice, but also in intensity. Thus, the increase in the practice of high-intensity physical activity and the alternation between sedentary and exercise periods involve an increase in inflammatory and acute painful episodes, being tendinitis and joint lesions the major problem, followed by sprains or bruises.

The pharmacological management of these conditions involves nonsteroidal anti-inflammatory drugs (NSAIDs), local corticosteroids, acetaminophen, chondroitin sulfate or even opioids. These are effective drugs but with serious side effects in some cases, especially in the long-term utilization. Severe drawbacks related to the prolonged utilization of these drugs include drug ineffectiveness, toxicity of certain agents, hypersensitivity, gastrointestinal hemorrhage, nauseas and even fatal outcomes including death and suicide. Importantly, increased abuse of painkillers has been reported in several countries, exceeding tobacco consumption and being considered a public health problem. Furthermore, the use of painkillers should be avoided in sensitive population groups including children and pregnant women, who are equally exposed to sustained or acute pain episodes.

Alternative solutions of greater safety but equivalent rapid relief and recovery effectiveness are a necessity. In this sense, the most useful approach are natural products, without tolerability concerns, compatible with other interventions and providing a rapid effect. These generalize access to effective treatment to both patients and physiotherapy professionals. Considering the well-established beneficial effects of physiotherapy in handling chronic pain, professionals need effective and safe solutions that they can use without concerns of side effects or pharmacological interactions, since they may not have access to the full medical record of the patients. In turn, the ability of handling self-treatment without concern increases the quality of life in patients suffering from pain-involving conditions.

This study evaluates the use of a topical cream composed by natural extracts with complementary and synergistic effects for pain management. Menthol reduces pain and increases blood flow, warming up the muscle and enhancing absorption of the rest of the extracts. Arnica montana reduces pain, has anti-inflammatory effects and potentiates tissue repair. Hypericum perforatum provides anti-inflammatory effect and drives tissue regeneration and scarring. Calendula officinalis reduces swelling and distension, boosts healing of mild injuries and prevents infection. Finally, Melaleuca alternifolia complements the anti-inflammatory effect and acts as a natural preservative due to its potent antimicrobial effect.

The synergistic combination of these natural ingredients may provide a convenient solution for the management acute or chronic pain. The aim of this study is to assess the benefits of the topical formulation in reducing musculoskeletal pain, both as an immediate relief of pain and as a solution for injury recovery.

ELIGIBILITY:
Inclusion Criteria:

* acute or chronic musculoskeletal pain scoring above 4 in the Visual Analogue Scale (VAS)
* diagnostic of either tendinopathy, vertebral algias, sprains or symptomatic osteoarthritis

Exclusion Criteria:

* diagnostic in either neuropathic chronic pain, fibromyalgia or neoplasia
* allergy to any ingredient in the formula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Average variation in pain at rest | 14 days (0, 7 and 14 days)
  pain reduction after intervention measured as per a Visual Analog Scale (1 - 10, higher values indicating more pain)
Average variation in pain in motion | 14 days (0, 7 and 14 days)
  pain reduction after intervention measured as per a Visual Analog Scale (1 - 10, higher values indicating more pain)

SECONDARY OUTCOMES:
Average variation in pain at rest | 2 hours (0, 30 minutes, 1 hour, 2 hours)
  pain reduction after intervention measured as per a Faces Scale (1 - 10, higher values indicating more pain)
Average variation in pain in motion | 2 hours (0, 30 minutes, 1 hour, 2 hours)
  pain reduction after intervention measured as per a Faces Scale (1 - 10, higher values indicating more pain)
Average variation in stiffness at rest | 2 hours (0, 30 minutes, 1 hour, 2 hours)
  stifness reduction after intervention measured as per a Stifness scale - (0) no stiffness, (1) slight stiffness, (2) moderate stiffness and (3) severe stiffness.
Average variation in stiffness in motion | 2 hours (0, 30 minutes, 1 hour, 2 hours)
  stifness reduction after intervention measured as per a Stifness scale - (0) no stiffness, (1) slight stiffness, (2) moderate stiffness and (3) severe stiffness.
Average variation in stiffness at rest | 14 days (0, 7 and 14 days)
  stifness reduction after intervention measured as per a Stifness scale -- (0) no stiffness, (1) slight stiffness, (2) moderate stiffness and (3) severe stiffness.
Average variation in stiffness in motion | 14 days (0, 7 and 14 days)
  stifness reduction after intervention measured as per a Stifness scale - (0) no stiffness, (1) slight stiffness, (2) moderate stiffness and (3) severe stiffness.
Recovery perception | 14 days (0, 7 and 14 days)
  Subjective perception of recovery as per a Likert scale ((1) meant fully recovered, (2) much better, (3) better, (4) same as before and (5) worse than before.)
Joint mobility | 14 days (0, 7 and 14 days)
  Joint mobility evaluation as per passive joint balance ((1) free mobility, (2) partial limitation, (3) moderate limitation and (4) severe limitation

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ramon, MD, PhD, Principal Investigator — Hospital QuiroSalud Barcelona
Locations (1):
- QuironSalud Hosiptal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No